CLINICAL TRIAL: NCT05351112
Title: Post-market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the Anatomical Shoulderᵀᴹ 2.0 Fracture System (Implants and Instrumentation) - A Retrospective and Prospective Consecutive Series Study
Brief Title: PMCF Study on the Safety, Performance and Clinical Benefits Data of the Anatomical Shoulder 2.0 Fracture System
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-44E
Record Dates: First submitted 2022-02-17; First posted 2022-04-28 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Proximal Humerus Fracture; Posttraumatic Arthrosis After Humeral Head Fracture; Posttraumatic Necrosis of the Humeral Head
Keywords: Post-Market Clinical Follow-Up Study; Medical Device; Performance; Safety; Clinical Benefits

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received the Anatomical Shoulder 2.0 Fracture: Anatomical Shoulder 2.0 Fracture

SUMMARY:
The study is a multicenter, retrospective and prospective, non-randomized, non-controlled and consecutive series post-market study. The purpose of this study is to collect long-term data confirming safety, performance and clinical benefits of the Anatomical Shoulder 2.0 Fracture System (Implants and Instrumentation) when used for fracture shoulder arthroplasty. The primary objective is the assessment of safety by analyzing implant survivorship. This will be established by recording the incidence and frequency of revisions, complications and adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified.

The secondary objective is the assessment of performance and clinical benefits by recording patient-reported clinical outcome measures (PROMs) as well as radiographic outcomes.

DETAILED DESCRIPTION:
The Anatomical Shoulder 2.0 Fracture System is intended for use in prosthetic replacement of the proximal humerus and the glenoid articular surface of the scapula during total, hemi and fracture shoulder arthroplasty. The system is intended for long-term implantation into the human shoulder joint to relieve pain and restore function in patients with adequate bone stock to support the prosthesis.

Two sites will be involved in this study. The aim is to include a total of 78 consecutive series cases who received the Anatomical Shoulder 2.0 Fracture starting from 2014. All potential study subjects will be required to participate in the Informed Consent Process.

Baseline data from the preop, intraop and immediate post-op intervals will be available in medical notes and collected retrospectively. During follow-up visits at 1, 3, 5, 7 and 10 years post-op (depending on patients' date of surgery), the patient will be asked to complete patient questionnaires. Moreover, a clinical assessment and a radiographic evaluation will be conducted. In addition, any complications and adverse events will also be collected during these follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older and skeletally mature
* Patients capable of understanding the surgeon's explanations and following his instructions, able and willing to participate in the follow-up program and who gave consent to take part in the study
* Replacement of the proximal humerus and the glenoid articular surface of the scapula during total-, hemi- and fracture shoulder arthroplasty in treatment of the following:

  1. Complex 3- and 4- part fractures of the proximal humerus with subluxation of the head fragment
  2. Complex 3- and 4- part fractures of the proximal humerus with loosening of the spongiosa in the head fragment
  3. Complex 3- and 4- part fractures of the proximal humerus with additional cross split of the head fragment
  4. Fracture instability after osteosynthesis of 3- and 4-part fracture fragments of the proximal humerus
  5. Posttraumatic necrosis of the humeral head
  6. Posttraumatic arthrosis after humeral head fracture

Exclusion Criteria:

* Patients who are unwilling or unable to give consent, not willing to return for study required follow-up visits and/or to comply with the follow-up program.
* The patient is known to be pregnant or breastfeeding
* Patients who have any condition that would in the judgment of the Investigator place the patient at undue risk or interfere with the study.
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, anticipated to be non-compliant).
* Patients with plans to relocate during the study follow-up period
* Signs of infection
* Extensive stiffening of the shoulder joint without pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of a consecutive series of cases implanted with the Anatomical Shoulder 2.0 Fracture System according to Zimmer Biomet's Instruction for Use (IFU) and who meet the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2034-01-21 (Estimated); Study Completion 2034-01-21 (Estimated)

PRIMARY OUTCOMES:
Incidence and frequency of revisions [Product safety based on implant survivorship] | 3-10 years
  Safety will be assessed by recording and analyzing the incidence and frequency of revisions, complications and adverse events. A Kaplan Meier survival curve will be calculated.

SECONDARY OUTCOMES:
Constant and Murley Score | 3-10 years
  The Constant and Murley score is a 100-point functional shoulder assessment tool in which higher scores reflect increased function. The subjective variables are pain (15 points) and function (activities of daily living - sleep, work, recreation/sport; 20 points), for a total of 35 points. The objective variables are active range of motion (clinician assessment; 40 points) and strength (25 points), for a total of 65 points.
Oxford Shoulder Score | 3-10 years
  The OSS is a self-assessment of shoulder pain and function with 12 items; pain (2), interference with pain (2), and daily functions (8). Each response is answered with a five point Likert scale. The total score is the sum of the 12 items, with lower scores indicating a more favorable outcome.
EuroQol Five Dimensions Questionnaire | 3-10 years
  The EQ-5D measures 5 dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with a total of 5 questions. It is accompanied by the patient's self-assessment with the VAS.
  Each dimension is assigned one of three discrete levels for evaluation on the day of administration:
  Level 1 - No problems, no disability Level 2 - Some problems, moderate disability Level 3 - A lot of problems, severe disability
  The final score is a five digit composite of the responses ranging between 33333 - 11111 with 243 possible combinations in between
X-rays | 3-10 years
  Performance and clinical benefits will be assessed by radiographic evaluation. Radiographs (A/P and axillary view) of the operated shoulder will be taken at each interval.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (1):
- Salamenca University Hospital, Salamanca, Spain